CLINICAL TRIAL: NCT06124274
Title: The Effect of Menstrual Phase and Oral Contraceptives on Muscle Protein Metabolism
Brief Title: Oral Contraceptive vs Menstrual Cycle Ex Vivo Model
Acronym: OCEV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OCEV
Record Dates: First submitted 2023-08-17; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Contraceptives, Oral; Sex Hormone
Keywords: Oral Contraceptive Use; Menstrual Cycle Phases; Protein Metabolism; Ex Vivo Model; Breath Test

STUDY DESIGN:
Intervention Model Description: This study uses a 4-way counterbalanced crossover design. A total 10 young women (Ages: 18-35 years old; 5 per OC and non-OC group) will be recruited and randomized to begin in either the mid-follicular (7-11 days after the onset of menses) or mid-luteal phase (5-9 days after ovulation) if part of non-OC group; and active pill (10-20 days within starting their new pill cycle) or withdrawal phase (at least 48hrs after their last pill) if part of the OC group. Participants of each group will take part in two metabolic trials, one in each phase of their menstrual cycle or pill cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mid-Follicular Phase (Experimental): 7-11 days after onset of menses.
  Interventions: Behavioral: Protein tracer drink
- Mid-Luteal Phase (Experimental): 5-9 days after ovulation (as confirmed with ovulation test kits).
  Interventions: Behavioral: Protein tracer drink
- Active pill phase (Experimental): 10-20 days after starting new pill cycle.
  Interventions: Behavioral: Protein tracer drink
- Withdrawal phase (Experimental): 48hrs after last pill (during placebo pill phase).
  Interventions: Behavioral: Protein tracer drink

INTERVENTIONS:
Behavioral: Protein tracer drink — Subjects will be fed a mixed-macronutrient beverage at rest (0.75g/kg lean body mass of carbohydrates; 0.125g/kg lean body mass of protein). Amino acid composition of the protein will be modelled off the composition of egg. Leucine content will be enriched to 5% with [13 Carbon(13C)]-leucine.

SUMMARY:
Despite comprising half the population, females are often left out of muscle research due to the impact of changing hormones during the menstrual cycle and when using oral contraceptives. This makes it hard to perform costly and invasive studies involving tracers to study muscle protein metabolism. Consequently, we lack a clear understanding of how these hormonal changes affect muscle growth.

There is a need for less invasive methods to study how sex hormones and oral contraceptives influence muscle protein metabolism. Ex vivo models, where serum from participants is applied to mouse muscle cell cultures, mimic the conditions of human muscle cells and can provide initial insights.

DETAILED DESCRIPTION:
The aim of the study is to develop a non-invasive model using serum from both oral contraceptive users and non-users at various stages of their cycles, to understand if different cycle or pill stages affect how muscles process proteins.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-29.9 kg/m2 (I.e., non-obese).
* For OC users: on monophasic OCs for > 3 months prior to study enrollment
* For non-OC users: regular menstrual cycles length (25-35 days) for at least 3 months prior to study and at least 6 months off of OCs.

Exclusion Criteria:

* Chronic disease diagnosis (cardiovascular, thyroid, diabetes)
* Current or recent remission of cancer
* Regular use of NSAID (except low-dose aspirin), anticoagulants
* Use of prescription drugs that would impact metabolism, e.g. Statins, Lithium, Attention-Deficit/Hyperactivity Disorder (ADHD) medication.
* Insertion of intrauterine device (IUD) - exception: copper
* Use of ergogenic aids such as creatine
* Regular Tabacco use
* Use of illicit drugs (growth hormones, testosterone)
* For non-OC users: Use of oral contraceptives for > 6 months prior to study enrollment - to ensure return to regular menstrual cycle.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Protein Synthesis (Murine Cell-Based Experiments, ex-vivo experiments) | 60 minutes
  Investigators will use human serum obtained from fasted and fed timepoints (-15, 20, 40 and 60 minutes following beverage consumption) to condition cell culture media (20% volume). To determine the effects of using fasted and/or fed 'human-conditioned' culture media on cell protein synthesis, puromycin incorporation (measure of protein synthesis) will be measured via western blot and expressed relative to a no-serum control. A two-way repeated measures ANOVA will be used to analyze outcomes with cycle stage and group (OC vs non-OC) used as factors

SECONDARY OUTCOMES:
Whole-body protein synthesis | 6 hours
  Investigators will measure the enrichment of [13 Carbon CO2 (13CO2)] in the breath by isotope ratio mass spectrometry (IRMS) in atom percent excess (APE). The measurement of carbon dioxide production (VCO2) and stable isotope tracer enrichment in the breath allows for the assessment of the rate at which amino acids are used for energy (i.e., oxidized), rather than for protein synthesis (i.e., retained in the body) by calculating the fraction of expired CO2 that contains 13C. Leucine retention (umol/kg) will then be calculated from the difference between the known amount of leucine provided (ingested) and leucine oxidation (as determined from 13CO2 breath enrichment).
Urinary Measures (Muscle Protein Breakdown) | 6 hours
  Investigators will measure urinary 3-methylhistidine (3MH) as an indirect marker of muscle protein breakdown over the course of the trial (6 hours) through pooled urine collection vs baseline urine.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Kortebi, PhD Student, Study Director — University of Toronto; Cassidy Tinline-Goodfellow, PhD (C), Study Director — University of Toronto; Jonathan Aguilera, PhD Student, Study Director — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No